CLINICAL TRIAL: NCT02112786
Title: Intermittent Versus Continuous Stimulation in Bilateral Sacral Neuromodulation for Overactive Bladder
Brief Title: Neuromodulation Implantation Settings Variation for Overactive Bladder
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: STIM-1; SUFU (Other: Society of Urodynamics, Female Pelvic Medicine & Urogenital Reconstruction (SUFU))
Record Dates: First submitted 2014-04-09; First posted 2014-04-14 (Estimated); Last update posted 2015-01-26 (Estimated); Status verified 2015-01

CONDITIONS: Overactive Bladder
Keywords: Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intermittent then Continuous (Active Comparator): This group will be set to intermittent stimulation first, then after the wash out period they will be switched to continuous stimulation.
  Interventions: Device: Intermittent or Continuous Setting RestorePrime Implanted Impulse Generator
- Continuous Then Intermitent (Active Comparator): This group will be set to continuous stimulation first, then switch to intermittent after the wash out time period.
  Interventions: Device: Intermittent or Continuous Setting RestorePrime Implanted Impulse Generator

INTERVENTIONS:
Device: Intermittent or Continuous Setting RestorePrime Implanted Impulse Generator — This is a routine procedure already performed, we are simply changing a post surgical setting to observe for improvement.
  Other Names: RestorePrime Implanted Impulse Generator

SUMMARY:
Participants receiving neuromodulation treatment for overactive bladder symptoms will be routinely fitted with an impulse generator. However, the setting on the impulse generator will be set to either intermittent or continuous stimulation. Participants will complete voiding logs and surveys for a month. Battery life will be interrogated.After a one week period were the device is turned off, the impulse generator will be turned to the opposite setting (intermittent or continuous) and the one month period will be repeated. Again, voiding logs, surveys, and battery life will be collected.

The purpose of this project is to investigate the outcomes of intermittent versus continuous stimulation in patients treated with sacral neuromodulation (SNM) for refractory overactive bladder (OAB) syndrome. In addition, the potential for an improved battery life with intermittent stimulation will be quantified.

DETAILED DESCRIPTION:
The objective of this project is to investigate the outcomes of intermittent versus continuous stimulation in patients treated with sacral neuromodulation (SNM) for refractory overactive bladder (OAB) syndrome. In addition, the potential for an improved battery life with intermittent stimulation will be quantified. Manufacturers recommended settings for newly implanted impulse generators (IPG); however, no standardized recommendations exist for further adjustments. Quality studies examining IPG parameters are lacking, partly due to the numerous setting variables, which can result in a multitude of permutations. When programming an IPG, an option for cycling simulation (16 seconds on, 8 seconds off) is available. It is theorized that because of a "carryover" effect, symptom relief will continue despite the stimulator being off. The potential benefit of the intermittent stimulation is an improved battery life, which may translate into a less frequent need for reimplantation with less morbidity. Participants receiving neuromodulation treatment for overactive bladder symptoms will be routinely fitted with an impulse generator in a pre-study phase. Patients who experience significant symptomatic improvement will receive a full bilateral sacral neuromodulator implantation and will be randomized to either intermittent or continuous stimulation. Participants will fill out voiding logs and surveys over a 12 week period. At that point, a one-week washout period during which the neuromodulator will be turned off. The impulse generator will then be turned to the alternate setting (intermittent or continuous) and the 12 week period will be repeated. Questionnaires and voiding diaries will be collected at each clinic visit. In total, subject participation will last approximately 25 weeks after full implantation of the bilateral leads and pulse generator.

ELIGIBILITY:
Inclusion criteria:

* patients age 18 to 85 with overactive bladder symptoms refractory to behavioral and anticholinergic therapy, detrusor overactivity on urodynamic study, surgically fit with ability to complete study forms, use patient programmer, and return for follow-up.

Patients must have attempted and failed noninvasive therapy for overactive bladder symptoms for at least 6 months prior to enrollment; previous treatments will be recorded. In addition, patients must be fluent in the English language to complete informed consent paperwork and study questionnaires.

Exclusion criteria:

* dementia,
* neurological conditions (spinal cord injury, multiple sclerosis),
* non-English speaking,
* acute urinary tract infection,
* primary pelvic pain,
* pregnancy or breast-feeding,
* urinary retention (postvoid residual greater than 100mL),
* history of bladder cancer in the past 5 years,
* history of nephrolithiasis or ureterolithiasis,
* anticoagulant therapy,
* implanted pacemaker/defibrillator, or
* anticipated need for future MRI.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-01; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Overactive Bladder Symptoms | Week 0, 2, 12, 13, 15, 25
  Symptom improvement with be tracked for overactive bladder symptoms through voiding logs and questionnaires.

SECONDARY OUTCOMES:
Battery Life | Week 0, 1, 12, 13, 15, 25
  Battery life of the implanted device will be interrogated at each follow up visit to measure longevity of battery.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Staack, MD, Phd, Principal Investigator — Loma LindaUniversity Medical Center
Locations (1):
- Loma Linda University Faculty Medical Offices, Loma Linda, California, United States

REFERENCES:
- [Background] Hu TW, Wagner TH, Bentkover JD, Leblanc K, Zhou SZ, Hunt T. Costs of urinary incontinence and overactive bladder in the United States: a comparative study. Urology. 2004 Mar;63(3):461-5. doi: 10.1016/j.urology.2003.10.037. PMID 15028438
- [Background] Nitti VW. Clinical impact of overactive bladder. Rev Urol. 2002;4 Suppl 4(Suppl 4):S2-6. PMID 16986018